CLINICAL TRIAL: NCT05862831
Title: Phase I Study to Evaluate the Tolerability, Safety, Pharmacokinetic and Primary Efficacy of PM1003 in Patients With Advanced Solid Tumors and Phase IIa Study to Evaluate the Primary Efficacy of PM1003 in Advanced Solid Tumors
Brief Title: Clinical Study of PM1003 in Phase I/IIa Treatment of Advanced Malignant Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biotheus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM1003-AB001M-ST-R
Record Dates: First submitted 2023-05-08; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Advanced Solid Tumors
Keywords: PD-L1, 4-1BB

STUDY DESIGN:
Intervention Model Description: In dose escalation stage, three subjects will be enrolled at the protocol starting dose of PM1032 for 21 Days DLT observation, followed by same dose every 2 weeks (Q2W) until they meet the discontinuation criteria.
  Dose escalation will proceed to the next dose level according to the 3+3 design.
  Dose expansion stage of the study will be initiated at the Sponsor's discretion at the dose level and treatment schedule which was established as the recommended Phase 2 dose (RP2D) in the dose escalation stage.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PM1003 (Experimental): PM1003 0.02mg/kg-10mg/kg
  Interventions: Biological: PM1003 Injection

INTERVENTIONS:
Biological: PM1003 Injection — Subjects will receive PM1003 by intravenous administration.

SUMMARY:
This is a single-arm, open-lable, multicenter phase I/IIa clinical trial evaluating the safety, tolerability, pharmacokinetics, and preliminary efficacy of PM1003 in the treatment of advanced solid tumors.

DETAILED DESCRIPTION:
PM1003 is a Bispecific Antibody Targeting PD-L1 and 4-1BB.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation in clinical study; fully understand the study and sign informed consent voluntarily; willing to follow and able to complete all test procedures;
2. Male or female aged 18 to 75 years;
3. Subjects with malignant tumor confirmed by histology or cytology;
4. Adequate organ function;
5. ECOG score was 0-1.
6. Pre-menopausal female subjects with negative blood pregnancy results within 7 days prior to the study treatment, and agree to abstain from sex or use medically approved effective contraceptive measures for 6 months from the date of signing the informed consent form to the end of the last medication;
7. Male subjects are agree to abstain from sex or use medically approved effective contraceptive methods for 6 months from the date of signing the informed consent form to the end of the last medication, and do not donate sperm during this period.

Exclusion Criteria:

1. History of severe allergic to macromolecular protein drugs, severe allergy to drugs or known allergy to any component of the drug in this study;
2. Treatment with any 4-1BB monoclonal antibody or 4-1BB-containing dual antibody immune co-stimulatory molecule agonist;
3. Current active infection requiring intravenous anti-infective therapy;
4. Current presence of uncontrolled pleural, pericardial, and peritoneal effusions;
5. Known history of alcohol abuse, psychotropic drug abuse or drug abuse;
6. History of neurological or psychiatric disorders, such as epilepsy, dementia, schizophrenia, etc.;
7. Anticipated need for any other form of antineoplastic drug treatment during the trial;
8. Women who are pregnant or breastfeeding;
9. Other conditions lead to inappropriate to participate in this study as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Estimated)
Dates: Start 2021-09-07 (Actual); Primary Completion 2025-09-07 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Dose Limited Toxicity（DLT） | up to 21 days
  Occurrence of DLT after receiving PM1003 injection
Assess the incidence and severity of treatment-related adverse events | Up to 30 days after last treatment
  The incidence and severity of treatment-emergent adverse events (TEAEs) and treatment related adverse events (TRAEs) graded according to NCI-CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Ye Guo, Principal Investigator — Shanghai Orient Hospital
Locations (2):
- China (2):
  - Cancer Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - Shanghai Orient Hospital, Shanghai